CLINICAL TRIAL: NCT04389359
Title: PROphylaxis for paTiEnts at Risk of COVID-19 infecTion (PROTECT): a Basket Trial of Prophylactic Interventions Amongst At-risk Patients
Brief Title: PROphylaxis for paTiEnts at Risk of COVID-19 infecTion
Acronym: PROTECT
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Regulatory approvals not received
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Thomas Hiemstra, Honorary Consultant Nephrologist, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A095590
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
Keywords: haemodialysis; transplant; immunosuppression; vasculitis; hydroxychloroquine; chemoprophylaxis; COVID-19
MeSH Terms: conditions — COVID-19; Vasculitis | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: PROTECT will use an innovative basket design to conduct a series of prospective, randomised comparisons in multiple vulnerable patient groups in the United Kingdom with the capabilities of assessing effects within specific patients groups, and across the pooled PROTECT cohort. Additional interventions may be added as these become available. Basket Trial design brings greater efficiency, due to running multiple comparisons within one master protocol. It also allows application of innovative Bayesian analysis methods that allow adaptive borrowing of information across populations. This will mean in the case that there is a consistent effect across populations, the trial will have greater power to find significant differences for individual patient groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCQ group (dialysis) (Experimental): Dialysis patients will receive Hydroxychloroquine sulfate 200 mg capsules or tablets (oral administration), as 600mg weekly in divided doses, given as 200mg after each dialysis session.
  Non-dialysis patients will receive Hydroxychloroquine sulfate, 400mg twice daily for two days, then 400mg weekly.
  Maximum treatment duration will be 26 weeks (6 months).
  Interventions: Drug: Hydroxychloroquine Sulfate 200 MG
- Control (No Intervention): Patients will continue with their usual medicines and clinical care without additional HCQ.

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate 200 MG — Hydroxychloroquine Sulfate administered orally for a maximum of 6 months. Doses population specific.
  Other Names: Plaquenil
  Arms: HCQ group (dialysis)

SUMMARY:
The PROTECT open-label randomised basket trial will assess the effectiveness of hydroxychloroquine (HCQ) as chemoprophylaxis against COVID-19 in multiple vulnerable populations in the United Kingdom.

DETAILED DESCRIPTION:
COVID-19 (novel coronavirus-induced disease) was declared a global pandemic by the WHO on 11th March 2020. Currently there are no drugs proven to treat or delay progression of COVID-19 and no vaccine is yet available. Efforts are underway to repurpose established drugs with well understood drug interactions and safety profiles. Vulnerable populations such as those receiving in-centre dialysis are largely excluded from ongoing trials.

The PROTECT Basket clinical trial aims to enrol patients at particularly high risk of COVID-19 and its complications, seeking to test treatments that either might prevent the disease from occurring or may reduce the number of cases where the disease becomes serious or life-threatening. The PROTECT trial will use innovative design and analysis methodologies to allow the simultaneous assessment of one or more treatments in multiple populations.

Patients will be eligible for recruitment to the trial if they fall within one of the following vulnerable populations: a) patients receiving in-centre haemodialysis, b) transplant patients, c) vasculitis, or d) other disease groups that may be added during the course of this trial.

PROTECT will use an innovate basket design to carry out a series of individually powered prospective, randomised comparisons in distinct vulnerable patient groups in the UK while applying Bayesian approaches to conduct pooled assessment of efficacy.

Once consented, eligible participants will be randomised to active treatment or control, stratified by PROTECT subpopulation (disease specific). Enrolment to the trial will be via an online platform and following informed consent subsequent assessments will be done via email or telephone thus reducing the burden to participants as well as reducing their exposure to COVID-19.

The master PROTECT protocol describes core components that are shared between disease specific appendices to the core protocol.

ELIGIBILITY:
Inclusion Criteria:

* Have no previous confirmed COVID-19 diagnosis
* Fall into one of the high risk population groups

Exclusion Criteria:

* Inability to provide informed consent
* Symptomatic for possible COVID-19 at baseline or symptoms highly suggestive of COVID-19 experienced since 1st March 2020
* Hypersensitivity reaction to hydroxychloroquine, chloroquine or 4-aminoquinolines or any formulation excipients
* Contraindication to taking hydroxychloroquine as prophylaxis e.g known epilepsy
* Already taking chloroquine, hydroxychloroquine or 4-aminoquinolines
* History of any retinopathy including diabetic retinopathy requiring laser therapy
* Taking medications which are contra-indicated alongside HCQ - Digoxin, Halofantrine, Amiodarone, Moxifloxacin, Cyclosporin, Mefloquine, Praziquantel, Tamoxifen
* Known history of prolonged QTc
* Type I diabetes or insulin-dependent type II diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Time to confirmed diagnosis of COVID-19 | To study completion, average 6 months
  The primary outcome for PROTECT is the time to confirmed COVID-19 infection from the date of randomisation. This will be captured via linkage with PHE or by direct reporting by sites.

SECONDARY OUTCOMES:
All-cause mortality | To study completion, average 6 months
  Death from any cause
Severity of COVID-19 disease | To study completion, average 6 months
  Severity will be assessed by requirement for hospitalisation, HDU/ICU admission or death and Length of inpatient stay.
Incidence of COVID-19 complications | To study completion, average 6 months
  Acute respiratory distress syndrome, viral pneumonitis, myocarditis/myocardial injury, acute kidney injury.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hiemstra, PhD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No